CLINICAL TRIAL: NCT00137670
Title: Effectiveness of a Video-based Educational Intervention to Prevent Human Immunodeficiency Virus (HIV) and Sexually Transmitted Diseases (STDs) Among Patients Attending STD Clinics
Brief Title: Video-based Intervention Study to Prevent HIV/Sexually Transmitted Diseases (STDs) Among STD Clinic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3500; R18/CCR921007; R18/CCR121005; R18/CCR821004
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Intervention studies; HIV
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Video-based HIV/STD prevention intervention

SUMMARY:
The purpose of this study is to assess the effectiveness of a brief 23-minute video-based educational waiting room intervention to reduce incident STD and high risk behavior among STD patients attending STD clinics in three United States (U.S.) cities.

DETAILED DESCRIPTION:
Approximately 15 million incident cases of sexually transmitted diseases (STDs) occur annually. As a result, primary prevention of HIV/STDs among persons who have chosen to be sexually active remains a high public health priority. A number of effective interventions to prevent HIV/STDs have been developed, however many require considerable time and resource investments from both service providers and participants. These programs are often difficult to implement and sustain over time. As a result, simple practical interventions that can reduce transmission or acquisition of HIV/STDs among STD clinic patients while being both easily implemented and sustainable are urgently needed, and will ultimately enhance the menu of effective programs that are currently available to the STD clinic population.

The intervention trial was designed to develop and evaluate a video-based HIV/STD prevention intervention for STD clinic clients. The primary goals of this study are to assess whether a brief video-based educational waiting room intervention can reduce STD incidence (STD incidence outcome study) and high risk behavior (behavioral outcome study) among male and female patients attending STD clinics, when compared with patients who receive standard clinic services. This study is being conducted as a multi-site trial in 3 urban STD clinics.

The intervention condition consists of a 23-minute educational video focused on preventing STD and HIV infection shown on a large television in the waiting room. Health promotion posters supplement the video. The control condition consists of the current standard waiting room experience in each city's STD clinic.

In the STD incidence outcome study, groups of patients attending the participating STD clinics are randomly assigned to blocks of clinic weeks to either the intervention or control condition. A waiver of informed consent was obtained whereby no subjects are actively enrolled for this phase of the study. Through a retrospective review of existing medical records and STD surveillance registry data, we will determine and compare the incidence of new STDs over a 12-month period (on average) by assigned waiting room conditions.

In the behavioral outcome study, investigators administer computer-based survey instruments to a random sample of ~1600 male and female patients (800 per arm) both at enrollment and at 3 months following their initial clinic visit. The primary objective of the behavioral study is to assess the effectiveness of the video intervention by comparing levels of high-risk behavior between waiting room conditions at 3 months' follow-up.

ELIGIBILITY:
Inclusion Criteria:

STD Incidence Outcome Study:

* All medical records for STD clinic patients visiting participating STD clinics during the study period.

Behavioral Outcome Study:

STD clinic patients:

* Not returning for a follow-up visit related to a previously diagnosed problem.
* 18 years of age or older.
* Not known to be HIV-infected by self-report.
* Able to understand and speak English fluently.
* Have not been previously seen as a patient in the clinic during an intervention block when the video was being played.
* Have never received a diagnosis of a condition that necessitates frequent return visits (e.g., genital warts) by self-report.
* Have not previously enrolled in the study.
* Reported being in the clinic waiting room at least 20 minutes.
* Do not plan to move outside the clinic's catchment area during the next 6 months.
* Are willing to provide informed consent for review of their medical record and STD surveillance registry information by study staff.
* Are not known to be pregnant according to self-report (women only).
* Are not known by clinicians or counselors to be seriously ill (e.g. new HIV diagnosis or severe pelvic inflammatory disease [PID]).
* Engaged in intercourse in the last three months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45000
Dates: Start 2002-04; Primary Completion 2006-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
STD Incidence Outcome Study: Compare STD incidence in groups by intervention and control conditions at 3, 6, and 12 months follow-up
Behavioral Outcome Study: Compare the incidence of risk behavior during the 3 month follow-up period among intervention and control conditions

SECONDARY OUTCOMES:
STD Incidence Outcome Study: Compare incidence of STD syndromes, and first episode of genital herpes or genital warts in intervention/control conditions
Behavioral Outcome Study: Compare additional measures of risk between intervention and control conditions at three months follow-up including potential mediators of risk and clinic utilization

CONTACTS AND LOCATIONS:
Overall Officials: Jeff D Klausner, MD, MPH, Principal Investigator — San Francisco Department of Public Health/ STD Prevention and Control Services; Cornelis A Rietmeijer, MD, PhD, Principal Investigator — Denver Public Health; Kevin Malotte, DrPH, Principal Investigator — California State University, Long Beach; Lydia N O'Donnell, Ed.D., Principal Investigator — Education Development Center, Inc.
Locations (4):
- United States (4):
  - California State University, Long Beach, Long Beach, California
  - San Francisco Department of Public Health, San Francisco, California
  - Denver Public Health, Denver, Colorado
  - Education Development Center, Inc., Newton, Massachusetts

REFERENCES:
- [Derived] Gallo MF, Margolis AD, Malotte CK, Rietmeijer CA, Klausner JD, O'Donnell L, Warner L; Safe in the City Study Group. Sexual abstinence and other behaviours immediately following a new STI diagnosis among STI clinic patients: Findings from the Safe in the City trial. Sex Transm Infect. 2016 May;92(3):206-10. doi: 10.1136/sextrans-2014-051982. Epub 2015 Dec 15. PMID 26670913
- [Derived] Warner L, Klausner JD, Rietmeijer CA, Malotte CK, O'Donnell L, Margolis AD, Greenwood GL, Richardson D, Vrungos S, O'Donnell CR, Borkowf CB; Safe in the City Study Group. Effect of a brief video intervention on incident infection among patients attending sexually transmitted disease clinics. PLoS Med. 2008 Jun 24;5(6):e135. doi: 10.1371/journal.pmed.0050135. PMID 18578564